CLINICAL TRIAL: NCT03305653
Title: Use of Esophageal String Test to Understand Symptoms, Inflammation, and Function in Eosinophilic Esophagitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Children's Hospital of Philadelphia (Other); Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17-0796
Record Dates: First submitted 2017-10-04; First posted 2017-10-10 (Actual); Results first posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Eosinophilic Esophagitis
Keywords: Pediatrics
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Current/historical diagnosis of EoE (Experimental): Subjects with current or historical diagnosis of EoE, or suspected of having EoE will complete the Esophageal String Test (EST) and EndoFLIP
  Interventions: Device: Esophageal String Test (EST)

INTERVENTIONS:
Device: Esophageal String Test (EST) — The EST is a gelatin capsule filled with a 90cm nylon string. A trailing end of the string protrudes from one end of the capsule. This end is taped to the cheek and the capsule is swallowed. As the capsule travels to the small intestine, the string inside the capsule is dislodged, leaving a string that goes from the cheek to the small intestine. The capsule dislodges from the string and the string is left in place, in the mouth, esophagus, stomach and small intestine for an hour. During this time, the string rubs against the inside of the esophagus and collects eosinophil proteins. After one hour, the string is removed through the mouth and placed in preservative to save the eosinophil proteins.

SUMMARY:
Presently, the only method available to monitor disease activity in Eosinophilic Esophagitis (EoE) is endoscopy with pathological review of biopsies. The overall goal of this study is to determine the ability of the Esophageal String Test (EST), a minimally invasive capsule based technology, to measure disease activity in children with EoE. Additionally, to determine esophageal distensibility in children presenting with EoE by using the EndoFLIP (functional luminal imaging probe) device during endoscopic procedures.

DETAILED DESCRIPTION:
When children are scheduled to undergo an endoscopy, research assistants will contact the family to arrange for the Esophageal String Test (EST) to be performed within one week of the endoscopy. The string test involves swallowing a small capsule with a thin piece of string inside it. The string unravels as the capsule goes down into the stomach. The investigator would tape the end of the string to the child's cheek, leaving it there for one hour. At the end of the hour, the investigator would remove the string by gently pulling it out through the mouth. Prior to swallowing the EST, the patient will complete the PEESS form (Pediatric Eosinophilic Esophagitis Symptom Scores) to assess symptoms.

The endoscopy and Endoscopic Reference System (EREFs) and EndoFLIP will be performed. The EndoFLIP is a slender probe covered by a smooth long balloon that is passed into the esophagus and slowly expanded with a salt solution. After standard of care endoscopic visualization, the FLIP, a 16 cm probe (Crospon) will be placed transorally and positioned 3 cm distal to the lower esophageal sphincter. Esophageal cross sectional areas and intrabag pressure will be measured during stepwise distensions beginning with 5 mL and increasing to a maximum of 70mL or intrabag pressure of 50 mmHg is achieved, whichever comes first. FLIP is FDA-approved without age restriction and its use has been approved by our IRBs previously. Primary results will be reported as distensibility plateau (mm).

Endoscopic severity: Endoscopic esophageal appearances will be scored using a validated EoE scoring system (EREFS). Five features of EoE will be scored: Edema (0-1), Rings (0-3) Exudates (0-2), Furrows (0-1), Stricture (0-1). Results will be reported as an inflammatory score (edema, exudates, furrows) and fibrostenotic score (rings, stricture). Functional Luminal Imaging Probe (FLIP):

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form.
* Willing to comply with all study procedures and be available for the duration of the study.
* Male or female, aged 7 to 18 years old, inclusive
* Undergoing upper Endoscopy with biopsy for clinical care at CHCO or CHOP
* Current or historical diagnosis of EoE, or suspected of having EoE

Exclusion Criteria:

* Known connective tissue disease, other eosinophilic disorders
* Past history of caustic injestion, esophageal surgery or other esophageal injury
* Known inflammatory bowel disease or esophageal motility disease (achalasia)
* Unwilling or unable to swallow the EST
* Oral or intravenous steroids in the preceding 60 days (not including swallowed topical fluticasone, budesonide, etc)
* Pregnancy
* Participation in a clinical study that may interfere with participation in this study

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Calies Menard-Katcher, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Current/Historical Diagnosis of EoE
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Current/Historical Diagnosis of EoE
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2
  Black | 2
  White | 15
  Hispanic | 2
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Eosinophilic Degranulating Protein Concentration
Description: Measure the concentration of eosinophilic degranulating protein on strings that have been swallowed by subjects diagnosed with EoE
Time Frame: Measurement at one hour, when string is removed
Population: Number of patients who completed swallowing the string
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Current/Historical Diagnosis of EoE
Number analyzed (Participants) | 20
ng/mL | 456.5 [6.6 to 3428.9]

ADVERSE EVENTS:
Time Frame: Up to 72 hours.
Arm/Group | Current/Historical Diagnosis of EoE
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-25): https://cdn.clinicaltrials.gov/large-docs/53/NCT03305653/Prot_SAP_000.pdf